CLINICAL TRIAL: NCT00386984
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Multicenter Phase III-Study to Evaluate the Efficacy of Octreotide in Patients With Inoperable Hepatocellular Carcinoma
Brief Title: Hector-Study to Evaluate the Efficacy of Octreotide in Patients With Inoperable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S 980916
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: hepatocellular carcinoma; Sandostatin-LAR; RCT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Somatostatin; Octreotide

INTERVENTIONS:
Drug: Somatostatin (octreotide)

SUMMARY:
A preliminary study has shown that the hormone-similar, growth-retarding drug octreotide can prolong survival time in patients with primary liver cancer. Due to methodological deficiencies of the preliminary study the results will be re-checked by the comparison of octreotide with an pseudo-drug (so-called placebo) primarily regarding to the survival time and secondarily concerning costs, side effects, patient cooperation and quality of life as well as specific conditions in the tumor tissue in both groups with 108 patients with primary liver cancer.

DETAILED DESCRIPTION:
A pilot study showed that octreotide can prolong survival time of patients with HCC. Due to methodological deficiencies the results of this pilot study will be re-evaluated by comparison of octreotide versus placebo primarily regarding to the global survival time and secondarily concerning the costs, side effects, patient compliance and quality of life as well as the Somatostatin receptors in the tumor tissue and its prognostic relevance in both groups with 108 patients with hepatocellular carcinoma.

An interim analysis was done after occurrence of the half of the events (deaths). No significant effect could be shown.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable patients
* histologically confirmed HCC or patients who refuse surgery and who otherwise (e.g. due to the advanced tumor stage) are not applicable for palliative local therapy (e.g. PEI, TACE, RFTA).
* Age: 18 years or older

Exclusion Criteria:

General:

* Patient with symptomatic Cholecyst-/Choledocholithiasis
* Patient with severe psychiatric disease.
* Participation in another clinical trial within the last 4 weeks.
* Simultaneous participation in another clinical examination.
* Legally incapacitated patient, who is not able, to understand nature, meaning and consequence of the study.
* Continuous drug or alcohol abuse.
* Patient with known HIV infection and antiretroviral therapy.
* Patient with not controllable infection disease.
* Pregnancy.

Study- and indication-specific exclusion criteria:

* Secondary malignant tumor without complete remission.
* Secondary malignant tumor with complete remission but current adjuvant therapy.
* Preliminary or current therapy with tamoxifen
* Pretreatment of the HCC.
* First-time diagnosis > 6 months before inclusion into the study.
* Severe hepatic encephalopathy, refractory to any treatment.
* Patients with operable HCC.
* Contraindication to i.m. injections.
* Hypersensitivity to octreotide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 1999-10; Study Completion 2003-02

PRIMARY OUTCOMES:
Overall survival time

SECONDARY OUTCOMES:
Costs of the treatment measured by days of in-patient treatment
Side effects
Patient compliance
Quality of life
Somatostatin receptors in the tumor tissue
Prognostic relevance of the Somatostatin receptors

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Allgaier, PD, Principal Investigator — Evangelischen Diakoniekrankenhaus
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Allgaier HP, Becker G, Blum HE. [A therapeutic study of hepatocellular carcinoma using octreotide (HECTOR). Hepatocellular Carcinoma: Treatment with Octreotide]. Dtsch Med Wochenschr. 2000 Mar 17;125(11):320. No abstract available. German. PMID 10761474